CLINICAL TRIAL: NCT01053598
Title: EVALUATION OF THE PERFORMANCE OF THE NITRATE REDUCTASE AND RESAZURIN TITRE ASSAY FOR THE DETECTION OF MYCOBACTERIUM TUBERCULOSIS COMPLEX FROM SPUTUM IN A HIGH TB AND HIV SETTING
Acronym: NRA RETA
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Mbarara University of Science and Technology (Other); Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: 821183
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Tuberculosis; HIV; AIDS; HIV Infections
Keywords: Mycobacterium tuberculosis; Nitrate Reductase Assay; NRA; REMA; RETA; Rezazurine
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Principle objective of this study is To evaluate the performance of NRA, NRA-p and REMA-p for the detection of M. tuberculosis complex from sputum samples from adult pulmonary TB suspects in a high TB and HIV prevalence setting, using LJ and MGIT culture as gold standard.

The Secondary objectives are:

* To measure the performance of each assay (NRA, NRA-p, REMA-p) in sputum smear-negative patients
* To describe the results of the colorimetric methods in HIV-positive and HIV-negative patients
* To assess the time to detection of both NRA/NRA-p, REMA-p methods.
* To evaluate the feasibility of the NRA, NRA-p, REMA-p methods.
* To determine the rate of contamination of the NRA, NRA-p and REMA-p assays.
* To evaluate the proportion and the clinical relevance of NTM among TB suspects in a high TB and HIV prevalence setting.
* To provide capacity building for TB diagnosis in Mbarara.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a leading cause of death in developing countries and its burden has been exacerbated by the concurrent HIV epidemic. Despite the advances in medicine, TB diagnosis still remains a challenge, especially in developing countries where diagnosis relies mostly on the detection of Mycobacterium tuberculosis complex (MTBC) by smear microscopy and/or culture. Smear microscopy is rapid, simple and not expensive but it lacks sensitivity. Culture on solid medium, which is performed in some well equipped laboratories, is more sensitive than microscopy but takes up to 8 weeks to obtain the result.

Colorimetric methods have been used for the rapid detection of drug sensitivity in M. tuberculosis either from isolates or directly from sputum. These methods rely on the detection of live bacteria through either enzymatic activity (nitrate reduction) or their ability to reduce an oxidation-reduction indicator, either in solid or liquid medium. They are fast, simple, and offer a good potential that should be evaluated for the diagnosis of TB.

The objective of this study is to evaluate the performance of colorimetric assays for the detection of M. tuberculosis complex from sputum samples from adult pulmonary TB suspects in a high TB and HIV prevalence setting, using Löwenstein Jensen (LJ) and Mycobacterium growth indicator tube (MGIT) culture as gold standard. The colorimetric methods evaluated here will be the solid medium-based nitrate reductase assay as described (NRA) or with an additional step using para Nitrobenzoic (PNB) acid for differentiation of MTBC and NTM (NRA-p), and the modified resazurin microplate assay, also using PNB for differentiation of MTBC and NTM (REMA-p).

. If any of the colorimetric assays is found to be accurate, significantly faster than conventional culture methods, and easy to perform, then it could be implemented in a tuberculosis culture laboratory. By reducing the time to detection compared to conventional culture and the costs compared to recent commercial methods, these assays offer a good alternative to conventional methods and might help to improve TB diagnosis in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary TB suspects as defined by a cough for more than 2 weeks
* Age 15 years and above
* Written informed consent signed

Exclusion Criteria:

* Producing pure blood sputum or clear saliva
* Producing less than 1 mL of sputum
* Receiving anti TB treatment (isoniazid, rifampicin, streptomycin, pyrazinamide, ethambutol) or quinolone for more than 1 week in the month before inclusion.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting at the outpatient department of the MRRH will be eligible if they meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of NRA, NRA-p and REMA-p for the detection of M. tuberculosis complex from sputum samples from adult pulmonary TB suspects in a high TB and HIV prevalence setting, using LJ and MGIT culture as gold standard | 7 Month

SECONDARY OUTCOMES:
-To measure the performance of each assay (NRA, NRA-p, REMA-p) in sputum smear-negative patients -To describe the results of the colorimetric methods in HIV-positive and HIV-negative patients | 7 Month

CONTACTS AND LOCATIONS:
Locations (1):
- Epicentre, Mbarara, Mbarara, Uganda